CLINICAL TRIAL: NCT07296211
Title: Increasing the Uptake of DSMES Program and Addressing Social Needs in Low-Income Vulnerable Immigrants
Acronym: INSPIRE
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: NYU Langone Health (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 24-01080; 5U48DP006778 (NIH)
Record Dates: First submitted 2025-12-09; First posted 2025-12-22 (Actual); Last update posted 2025-12-22 (Actual); Status verified 2025-12

CONDITIONS: Type2 Diabetes Mellitus
Keywords: T2DM; Diabetes
MeSH Terms: conditions — Diabetes Mellitus | interventions — Telemedicine; Palliative Care; Videotape Recording

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Patients in a CHW-enabled clinic that receive mobile health (mHealth) videos (Experimental): For the first 6 months participants will receive CHW-enabled services from their clinic. Over the next 6 months participants will receive 24 culturally tailored diabetes education videos via text message.
  Interventions: Behavioral: CHW-enabled CCL; Behavioral: Mobile health (mHealth) diabetes self-management education and support (DSMES) videos
- Patients in a CHW-enabled clinic that do not receive mHealth videos (Experimental): For the first 6 months participants will receive CHW-enabled services from their clinic. Over the next 6 months participants will continue to receive standard of care (SOC).
  Interventions: Behavioral: CHW-enabled CCL
- Patients in a standard clinic that do not receive mHealth videos (No Intervention): For 12 months participants will be followed as they receive SOC from their clinic.

INTERVENTIONS:
Behavioral: CHW-enabled CCL — The FHCs has access to the CHW-enabled CCL. With this intervention, participants will be screened for social determinants of health (SDoH) and be referred to care and social services that address any identified needs.
  Arms: Patients in a CHW-enabled clinic that do not receive mHealth videos; Patients in a CHW-enabled clinic that receive mobile health (mHealth) videos
Behavioral: Mobile health (mHealth) diabetes self-management education and support (DSMES) videos — Participants will receive 24 culturally tailored DSMES videos through text message.
  Arms: Patients in a CHW-enabled clinic that receive mobile health (mHealth) videos

SUMMARY:
The purpose of this study is to evaluate a multi-level approach to improve diabetes control via access to social service supports and online, culturally-tailored diabetes self-management education and support (DSMES) videos among a community of primarily Chinese and Latino/a immigrants. The study aims to assess patient uptake, provider adoption, and INSPIRE program acceptability, appropriateness, feasibility, fidelity, penetration/reach, and maintenance.

DETAILED DESCRIPTION:
In stage 1, the 8 family health center (FHC) clinics will be randomized 1:1 into Experimental Cohort A, which will receive the Community Health Worker (CHW)-enabled community-clinic linkage model (CCL) or Control Cohort B, with FHCs that will not receive the CHW-enabled CCL. Then, in stage 2, patients in clinics that received the CHW-enabled CCL will be randomized in a 1:1 ratio to Arm A who will receive text-based mhealth diabetes education videos or Arm B who will not receive mhealth.

ELIGIBILITY:
Inclusion Criteria:

To be eligible to participate in this study, the patient participant must meet all the following criteria:

1. ≥18 years old and ≤ 70 years old
2. Self-identify their primary language as English, Mandarin, Cantonese, or Spanish
3. Diagnosed with T2DM
4. Has their most recent HbA1c ≥8% or have a new diagnosis of T2DM within the past 6 months

For patient participants randomized to the mHealth cohort, they must meet the below inclusion criteria

1. Willing to receive text messages with brief videos regarding T2DM management

Exclusion Criteria:

1. Unable or unwilling to provide informed consent
2. Unable to participate meaningfully in the intervention (e.g. uncorrected sight and hearing impairment)
3. Is currently pregnant (Pregnant women will be excluded from this study because they may have special dietary restrictions that are not covered by our DSMES videos for the general population with T2DM.)

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 480 (Estimated)
Dates: Start 2026-01 (Estimated); Primary Completion 2028-12 (Estimated); Study Completion 2029-06 (Estimated)

PRIMARY OUTCOMES:
Change in HbA1c levels | Baseline, Month 6

SECONDARY OUTCOMES:
Level of satisfaction with community-clinic linkage (CCL) and mHealth | Month 12
  Participants are asked to rate satisfaction on a scale of 1 (not satisfied at all) to 10 (very satisfied).
Percentage of patients accepting Community Health Worker (CHW) support | Month 12
Percentage of patients accepting mHealth | Month 12
Percent completion of social service referrals | Month 6
Percent mhealth videos watched | Month 12

CONTACTS AND LOCATIONS:
Overall Officials: Nadia Islam, PhD, Principal Investigator — NYU Langone Health
Locations (1):
- NYU Langone Health, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
The de-identified participant data from the final research dataset will be shared upon reasonable request beginning 9 to 36 months after publication or as required by a condition of awards or supporting agreements, provided the requesting investigator executes a data use agreement with NYU Langone Health. This instance of data sharing will also require separate IRB review as well as review from NYU Langone's Data Sharing Strategy Board (DSSB). Requests should be directed to: Brita.Roy@nyulangone.org. The protocol and statistical analysis plan will be posted on Clinicaltrials.gov only as required by federal regulation or supporting awards and agreements.
Supporting Information: Study Protocol, SAP
Time Frame: Beginning 9 months and ending 36 months following article publication or as required by a condition of awards and agreements supporting the research.
Access Criteria: The investigator who proposed to use the data will be granted access upon reasonable request. Requests should be directed to Brita.Roy@nyulangone.org. To gain access, data requestors will need to sign a data access agreement. This instance of data sharing will also require separate IRB review as well as review from NYU Langone's DSSB.